CLINICAL TRIAL: NCT01189435
Title: A Phase 2 Trial of Erlotinib Re-Challenge for Recurrent EGFR-mutant Lung Cancer in Patients Who Previously Received Adjuvant Erlotinib or Gefitinib
Brief Title: Erlotinib Re-Challenge for Recurrent EGFR-mutant Lung Cancer in Patients Who Previously Received Adjuvant Erlotinib or Gefitinib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-097
Record Dates: First submitted 2010-08-25; First posted 2010-08-26 (Estimated); Results first posted 2015-04-21 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-10

CONDITIONS: Lung Cancer
Keywords: OSI-774, TARCEVA (ERLOTINIB); Lung; recurrent; 10-097; Gefitinib
MeSH Terms: conditions — Lung Neoplasms; Recurrence | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- erlotinib (Experimental): This will be a single institution, single-arm, two-stage, open-label study of erlotinib in the treatment of patients with recurrent EGFR-mutant lung cancer following completion of adjuvant erlotinib or gefitinib therapy.
  Interventions: Drug: erlotinib

INTERVENTIONS:
Drug: erlotinib — After baseline evaluation, patients will initiate treatment with erlotinib 150 mg daily, or at maximum previous tolerated dose. Initial response assessment will be done during the fourth week of therapy, during the eighth week of therapy, and then every 8 weeks thereafter. Patients will continue on therapy until disease progression by RECIST.

SUMMARY:
The purpose of this study is to measure the ability of erlotinib to effectively treat recurrent lung cancer which carries an EGFR mutation lung cancer after prior treatment with erlotinib or gefitinib received in the post-surgical or post-radiation setting.

ELIGIBILITY:
Inclusion Criteria:

* A history of stage I-IIIB NSCLC
* Previously underdone definitive surgery or radiation
* Received prior adjuvant treatment or neoadjuvant with erlotinib or gefitinib for a total of at least 3 months at any time
* Stopped adjuvant erlotinib or neoadjuvant at least 2 months prior to date of first imaging demonstrating recurrence
* Pathologic evidence of recurrent lung cancer, confirmed at MSKCC EGFR sensitizing mutation (point mutation in exons 18 or 21, or deletion in exon 19) must be documented in the primary or recurrent tumor
* Tissue from their recurrent tumor must be submitted for EGFR mutation testing, and to evaluate for the presence of the T790M mutation (results do not need to have been reported to be eligible)
* Measurable disease by RECIST; if received prior irradiation, then must have a target lesion outside the irradiated field
* Signed informed consent
* Age > or = to 21 years old
* Persons of reproductive potential must agree to use an adequate method of contraception throughout treatment and for at least 4 weeks after study drug is stopped

Exclusion Criteria:

* Prior progressive disease while receiving erlotinib or gefitinib therapy
* Patients with known pre-existing interstitial lung disease
* Total bilirubin greater than 1.8 mg/dl, excepting patients known to have Gilbert's syndrome
* AST or ALT greater than five times the upper limit of normal
* Pregnant or lactating women
* Medically unfit for erlotinib therapy as determined by treating oncologist

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Azzoli, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erlotinib
Started | 2
Completed | 0
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: To Examine the Objective Response Rate (ORR) of Single-agent Erlotinib
Description: in recurrent EGFR-mutant lung cancer, given to patients who previously received adjuvant erlotinib or gefitinib
Time Frame: 2 years
Arm/Group | Erlotinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Erlotinib
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib (N=2)
Bilirubin (hyperbilirubinemia) (Blood and lymphatic system disorders) | 1 (1)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes